CLINICAL TRIAL: NCT03292016
Title: A Comparative Bioavailability Study to Evaluate the Single Dose Pharmacokinetic Properties of APL-130277 With Two Different Formulations of Subcutaneous Apomorphine in a Randomized, 3-Period Crossover Design in Subjects With Parkinson's Disease Complicated by Motor Fluctuations ("OFF" Episodes)
Brief Title: A Study That Compares the Extent to Which Apomorphine Becomes Available in the Body After Taking Either an Investigational Drug Containing Apomorphine or Apomorphine That is Injected Under the Skin in People With PD Complicated by "OFF" Episodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTH-203
Record Dates: First submitted 2017-09-11; First posted 2017-09-25 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease
Keywords: Off Episodes; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- APL-130277, sublingual thin film (Experimental): APL-130277, sublingual thin film, once daily
  Interventions: Drug: APL-130277
- Subcutaneous APO-go (Active Comparator): Subcutaneous APO-go, once daily
  Interventions: Drug: APO-go
- Subcutaneous APOKYN (Active Comparator): Subcutaneous APOKYN, once daily
  Interventions: Drug: Apokyn

INTERVENTIONS:
Drug: APL-130277 — APL-130277 sublingual thin film
  Other Names: amomorphine
  Arms: APL-130277, sublingual thin film
Drug: APO-go — Subcutaneous APO-go
  Other Names: amomorphine
  Arms: Subcutaneous APO-go
Drug: Apokyn — Subcutaneous APOKYN
  Other Names: amomorphine
  Arms: Subcutaneous APOKYN

SUMMARY:
A study that compares the extent to which apomorphine becomes available in the body after taking either an investigational drug containing apomorphine or apomorphine that is injected under the skin in people with PD complicated by "OFF" episodes.

DETAILED DESCRIPTION:
This multi-center study will aim to evaluate the pharmacokinetics (PK) and comparative bioavailability of a single dose of APL-130277 sublingual thin film with subcutaneous (s.c.) APO-go® and s.c. APOKYN® in subjects with Parkinson's disease (PD). The dose of APOKYN® (≤ 5 mg) will be based on the subjects' current prescribed dose. The study is designed as an open-label, randomized, three-way crossover. Subjects will receive all three treatment arms with a minimum 1-day wash-out between each visit (excluding the screening visit) and will be randomly assigned to one of the six sequences

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Clinical diagnosis of Idiopathic PD, consistent with UK Brain Bank Criteria (excluding the "more than one affected relative" criterion).
3. Clinically meaningful response to Levodopa (L-Dopa) with well-defined "OFF" episodes, as determined by the Investigator.
4. Receiving APOKYN® of ≤ 5 mg per dose for at least 4 weeks before the Screening Visit.
5. Receiving stable doses of L-Dopa/carbidopa (immediate or sustained release) administered at least 4 times per day OR Rytary™ administered 3 times per day, for at least 4 weeks before the Screening Visit. Adjunctive PD medication regimens must be maintained at a stable dose for at least 4 weeks prior to the Screening Visit with the exception that MAOB inhibitors must be maintained at a stable level for at least 8 weeks prior to the Screening Visit.
6. No planned medication change(s) or surgical intervention anticipated during the course of study.
7. Patients must experience a well-defined "OFF" episode in the morning if they do not take their morning PD medications on schedule, and must be willing to delay morning doses on the 3 study dosing days
8. Stage III or less on the modified Hoehn and Yahr scale in the "ON" state.
9. Mini-Mental State Examination (MMSE) score > 23.
10. If female and of childbearing potential, must agree to use one of the following methods of birth control:

    * Oral contraceptive;
    * Contraceptive patch;
    * Barrier (diaphragm, sponge or condom) plus spermicidal preparations;
    * Intrauterine contraceptive system;
    * Levonorgestrel implant;
    * Medroxyprogesterone acetate contraceptive injection;
    * Complete abstinence from sexual intercourse;
    * Hormonal vaginal contraceptive ring; or
    * Surgical sterilization or partner sterile (must have documented proof).
11. Male patients must be either surgically sterile, agree to be sexually abstinent or use a barrier method of birth control (e.g., condom) or maintain a monogamous relationship with a person who is not of child-bearing potential from first study drug administration until 30days after final drug administration.
12. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures to complete the study.
13. Able to understand the consent form, and to provide written informed consent

Exclusion Criteria:

1. Atypical or secondary parkinsonism.
2. Previous treatment with any of the following: continuous subcutaneous (s.c.) apomorphine infusion; or Duodopa/Duopa.
3. Contraindications to APO-go® or APOKYN® or hypersensitivity to apomorphine hydrochloride or any marcrolide antibiotic or any of the ingredients APO-go® or APOKYN® (notably sodium metabisulfite).
4. Female who is pregnant or lactating.
5. Participation in a clinical trial within 30 days prior to the Screening Visit.
6. Receipt of any investigational (ie, unapproved) medication within 30 days prior to the Screening Visit.
7. Any selective 5HT3 antagonists (ie, ondansetron, granisetron, dolasetron, palonosetron, alosetron), dopamine antagonists (excluding quetiapine and clozapine) or dopamine depleting agents within 30 days prior to the Screening Visit.
8. Drug or alcohol dependency in the past 12 months.
9. History of malignant melanoma.
10. Clinically significant medical, surgical, or laboratory abnormality in the opinion of the Investigator.
11. Major psychiatric disorder including, but not limited to, dementia, bipolar disorder, psychosis, or any disorder that, in the opinion of the Investigator, requires ongoing treatment that would make study participation unsafe or make treatment compliance difficult.
12. History of clinically significant hallucinations during the past 6 months.
13. History of clinically significant impulse control disorder(s).
14. Dementia that precludes providing informed consent or would interfere with participation in the study.
15. Current suicidal ideation within one year prior to the Screening Visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) or attempted suicide within the last 5 years.
16. Donation of blood plasma in the 30 days prior to first dosing.
17. Cankers or mouth sores within 30 days prior to the Screening Visit, or other clinically significant oral pathology in the opinion of the Investigator. The Investigator should follow-up with an appropriate specialist on any finding, if indicated, before enrolling a patient into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Mecdical Director, Study Chair — Sunovion Pharmacetuicals Inc.
Locations (3):
- United States (3):
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Parkinson's Disese Treatment Center of SW Florida, Port Charlotte, Florida
  - QUEST Research Institute, Farmington Hills, Michigan

REFERENCES:
- [Derived] Agbo F, Isaacson SH, Gil R, Chiu YY, Brantley SJ, Bhargava P, Navia B. Pharmacokinetics and Comparative Bioavailability of Apomorphine Sublingual Film and Subcutaneous Apomorphine Formulations in Patients with Parkinson's Disease and "OFF" Episodes: Results of a Randomized, Three-Way Crossover, Open-Label Study. Neurol Ther. 2021 Dec;10(2):693-709. doi: 10.1007/s40120-021-00251-6. Epub 2021 May 15. PMID 33991326

RESULTS

PARTICIPANT FLOW:
Groups:
- APL-130277, Then APOKYN, Then APO-go: Sequence 1: Participants first received APL-130277 (approximate equivalent dose to current APOKYN dose: 15 mg/ 20 mg/ 25 mg/ 30 mg) in the 'OFF' state. After a washout period of at least one day, they received APOKYN (current prescribed dose : 2 mg/3 mg/4mg/5 mg) in the 'OFF' state. After a washout period of at least one day, they received APO-go ( same dose as APOKYN: 2 mg/3 mg/4mg/5 mg) in the 'OFF' state.
- APL-130277, Then APO-go, Then APOKYN: Sequence 2: Participants first received APL-130277 (approximate equivalent dose to current APOKYN dose: 15 mg/ 20 mg/ 25 mg/ 30 mg) in the 'OFF' state. After a washout period of at least one day, they received APO-go (same dose as APOKYN 2 mg/3 mg/4mg/5 mg) in the 'OFF' state. After a washout period of at least one day, they received APOKYN (current prescribed dose : 2 mg/3 mg/4mg/5 mg) in the 'OFF' state.
- APOKYN, Then APL-130277, Then APO-go: Sequence 3: Participants first received APOKYN (current prescribed dose : 2 mg/3 mg/4mg/5 mg) in the 'OFF' state. After a washout period of at least one day, they received APL-130277 (approximate equivalent dose to current APOKYN dose: 15 mg/ 20 mg/ 25 mg/ 30 mg) in the 'OFF' state. After a washout period of at least one day, they received APO-go (same dose as APOKYN 2 mg/3 mg/4mg/5 mg) in the 'OFF' state.
- APOKYN, Then APO-go, Then APL-130277: Sequence 4: Participants first received APOKYN (current prescribed dose : 2 mg/3 mg/4mg/5 mg) in the 'OFF' state. After a washout period of at least one day, they received APO-go (same dose as APOKYN 2 mg/3 mg/4mg/5 mg) in the 'OFF' state. After a washout period of at least one day, they received APL-130277 (approximate equivalent dose to current APOKYN dose: 15 mg/ 20 mg/ 25 mg/ 30 mg) in the 'OFF' state.
- APO-go, Then APL-130277, Then APOKYN: Sequence 5: Participants first received APO-go (same dose as APOKYN 2 mg/3 mg/4mg/5 mg) in the 'OFF' state. After a washout period of at least one day, they received APL-130277 (approximate equivalent dose to current APOKYN dose: 15 mg/ 20 mg/ 25 mg/ 30 mg) in the 'OFF' state. After a washout period of at least one day, they received APOKYN (current prescribed dose : 2 mg/3 mg/4mg/5 mg) in the 'OFF' state.
- APO-go, Then APOKYN, Then APL-130277: Sequence 6: Participants first received APO-go (same dose as APOKYN 2 mg/3 mg/4mg/5 mg) in the 'OFF' state. After a washout period of at least one day, they received APOKYN (current prescribed dose : 2 mg/3 mg/4mg/5 mg) in the 'OFF' state. After a washout period of at least one day, they received APL-130277 (approximate equivalent dose to current APOKYN dose: 15 mg/ 20 mg/ 25 mg/ 30 mg) in the 'OFF' state.
Period: First Intervention
Arm/Group | APL-130277, Then APOKYN, Then APO-go | APL-130277, Then APO-go, Then APOKYN | APOKYN, Then APL-130277, Then APO-go | APOKYN, Then APO-go, Then APL-130277 | APO-go, Then APL-130277, Then APOKYN | APO-go, Then APOKYN, Then APL-130277
Started | 1 | 1 | 2 | 1 | 1 | 2
Completed | 1 | 1 | 2 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout
Arm/Group | APL-130277, Then APOKYN, Then APO-go | APL-130277, Then APO-go, Then APOKYN | APOKYN, Then APL-130277, Then APO-go | APOKYN, Then APO-go, Then APL-130277 | APO-go, Then APL-130277, Then APOKYN | APO-go, Then APOKYN, Then APL-130277
Started | 1 | 1 | 2 | 1 | 1 | 2
Completed | 1 | 1 | 2 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | APL-130277, Then APOKYN, Then APO-go | APL-130277, Then APO-go, Then APOKYN | APOKYN, Then APL-130277, Then APO-go | APOKYN, Then APO-go, Then APL-130277 | APO-go, Then APL-130277, Then APOKYN | APO-go, Then APOKYN, Then APL-130277
Started | 1 | 1 | 2 | 1 | 1 | 2
Completed | 1 | 1 | 2 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout
Arm/Group | APL-130277, Then APOKYN, Then APO-go | APL-130277, Then APO-go, Then APOKYN | APOKYN, Then APL-130277, Then APO-go | APOKYN, Then APO-go, Then APL-130277 | APO-go, Then APL-130277, Then APOKYN | APO-go, Then APOKYN, Then APL-130277
Started | 1 | 1 | 2 | 1 | 1 | 2
Completed | 1 | 0 | 2 | 1 | 1 | 2
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | APL-130277, Then APOKYN, Then APO-go | APL-130277, Then APO-go, Then APOKYN | APOKYN, Then APL-130277, Then APO-go | APOKYN, Then APO-go, Then APL-130277 | APO-go, Then APL-130277, Then APOKYN | APO-go, Then APOKYN, Then APL-130277
Started | 1 | 0 | 2 | 1 | 1 | 2
Completed | 1 | 0 | 2 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APL-130277, Then APOKYN, Then APO-go | APL-130277, Then APO-go, Then APOKYN | APOKYN, Then APL-130277, Then APO-go | APOKYN, Then APO-go, Then APL-130277 | APO-go, Then APL-130277, Then APOKYN | APO-go, Then APOKYN, Then APL-130277 | Total
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 1 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 0 | 0 | 1 | 3
  >=65 years | 1 | 0 | 1 | 1 | 1 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75 | 51 | 67.5 (9.19) | 67 | 73 | 68.5 (9.19) | 67.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Male | 1 | 0 | 2 | 1 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2 | 1 | 1 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 2 | 1 | 1 | 2 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Country [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2 | 1 | 1 | 2 | 8
Height (cm) at Baseline [Mean (Standard Deviation); unit: cm] | 172.7 | 157.5 | 174.95 (11.243) | 175.3 | 177.8 | 171.25 (19.445) | 171.96 (10.545)
Body Weight (kg) at Baseline [Mean (Standard Deviation); unit: kg] | 86.3 | 59.4 | 86.7 (20.506) | 73 | 84.4 | 71.2 (25.032) | 77.36 (15.895)
BMI (kg/m2) at Baseline [Mean (Standard Deviation); unit: kg/m^2] | 28.9 | 23.9 | 28.1 (3.111) | 23.8 | 26.7 | 23.8 (3.111) | 25.89 (2.826)
ON State Mod. Hoehn & Yahr Score [Mean (Standard Deviation); unit: Score] — The modified Hoehn and Yahr Scale (HYS) provides a global assessment of severity in Parkinson's Disease based on clinical findings and functional disability.•Stage 0:(No signs of disease, through Stage 5: Wheelchair bound or bedridden unless aided.
  Higher rates describe an increase severity of the disease.
  Score | 2 | 2 | 2.5 (0) | 2.5 | 3 | 2.5 (0.707) | 2.44 (0.417)
Mini-Mental Status Total Score [Mean (Standard Deviation); unit: Score] — Mini-Mental State Examination (MMSE) is used to evaluate a person's cognitive and mental function. Score range is 0-30 with lower scores showing higher impairment.
  Score | 30 | 30 | 26.5 (2.12) | 25 | 27 | 27.5 (3.54) | 27.5 (2.33)
Child-bearing potential [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 0 | 0 | 0 | 0 | 1
  No | 0 | 0 | 0 | 0 | 0 | 1 | 1
  N/A | 1 | 0 | 2 | 1 | 1 | 1 | 6
Smoking Status [Count of Participants; unit: Participants]
  Has never smoked | 1 | 1 | 0 | 1 | 1 | 2 | 6
  Former Smoker | 0 | 0 | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Dose normalized maximum observed plasma concentration (Cmax)
Time Frame: Day 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: (ng/mL)/(mg)
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 7 | 8
(ng/mL)/(mg) | 0.281 [0.191 to 0.413] | 2.29 [1.46 to 3.59] | 2.74 [1.82 to 4.13]
Statistical Analysis 1: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Sample size of 12 subjects, a two-sided 90% CI for the difference in paired PK parameter means on the log scale will have an interval that extends no more than 0.221 units from the observed difference with 90% coverage probability. Assumes CV of 35% for the difference on the original scale; Test type: Other; Mixed Models Analysis; With fixed effects-treatment and period, random effect-subject nested within sequence to analyze natural-log transformed dose normalized parameter; Geometric Mean ratio (APL-130277/APOKYN) = 12.3, 90% CI 2-sided [7.5 to 20.3]
Statistical Analysis 2: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Geometric Mean ratio (APL-130277/APO-go) = 10.3, 90% CI 2-sided [6.5 to 16.3]
Statistical Analysis 3: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other — relative bioavailibilty; Geometric Mean ratio (APOKYN/APO-go) = 83.4, 90% CI 2-sided [50.5 to 137.6]
Statistical Analysis 4: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Ratio = 0.21 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 20 mg and APO-Go 3 mg
Statistical Analysis 5: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; Ratio = 0.13 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 20 mg and APOKYN 3 mg
Statistical Analysis 6: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; Ratio = 1.16 — The comparative bioavailability calculated as the ratio of the Test/Reference between APO-Go 3 mg and APOKYN 3 mg
Statistical Analysis 7: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Ratio = 0.16 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 25 mg and APO-Go 4 mg
Statistical Analysis 8: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; Ratio = 0.17 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 25 mg and APOKYN 4 mg
Statistical Analysis 9: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; Ratio = 1.12 — The comparative bioavailability calculated as the ratio of the Test/Reference between APO-Go 4 mg and APOKYN 4 mg
Statistical Analysis 10: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Ratio = 0.08 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 30 mg and APO-Go 5 mg
Statistical Analysis 11: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; Ratio = 0.09 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 30 mg and APOKYN 5 mg
Statistical Analysis 12: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; Ratio = 1.04 — The comparative bioavailability calculated as the ratio of the Test/Reference between APO-Go 5 mg and APOKYN 5 mg

2. Primary Outcome: Observed Time of the Maximum Concentration (Tmax)
Description: Time from dosing to Cmax, observed by inspection of individual subject plots of plasma concentration versus time.
Time Frame: Day 1
Population: Tmax summary statistics were summarized by dose levels and the inferential statistics was done across all dose levels.
Measure: Median (Full Range); unit: hour
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 7 | 8
hour
  APL 20 mg, APOKYN 3 mg, and APO-go 3 mg: number analyzed (Participants) | 3 | 2 | 2
  APL 20 mg, APOKYN 3 mg, and APO-go 3 mg | 0.75 [0.52 to 0.75] | 0.38 [0.25 to 0.50] | 0.38 [0.25 to 0.50]
  APL 25 mg, APOKYN 4 mg, and APO-go 4 mg: number analyzed (Participants) | 2 | 2 | 2
  APL 25 mg, APOKYN 4 mg, and APO-go 4 mg | 0.63 [0.25 to 1.02] | 0.25 [0.25 to 0.25] | 0.26 [0.25 to 0.27]
  APL 30 mg, APOKYN 5 mg, and APO-go 5 mg: number analyzed (Participants) | 3 | 2 | 3
  APL 30 mg, APOKYN 5 mg, and APO-go 5 mg | 0.75 [0.50 to 1.00] | 0.38 [0.25 to 0.50] | 0.25 [0.25 to 0.50]
Statistical Analysis 1: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; p = 0.0625, Sign test
Statistical Analysis 2: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; p = 0.0313, Sign test
Statistical Analysis 3: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; p > 0.9999, Sign test

3. Primary Outcome: Area Under the Concentration- Time Curve (AUC Last)
Description: area under the concentration-time curve from time zero to the last measurable plasma concentration-time curve using the linear up log down trapezoidal rule.
Time Frame: Day 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: (hxng/mL)/(mg)
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 7 | 8
(hxng/mL)/(mg) | 0.500 [0.344 to 0.726] | 2.91 [1.97 to 4.30] | 3.00 [2.05 to 4.39]
Statistical Analysis 1: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio (APL-130277/APOKYN) = 17.2, 90% CI 2-sided [13.1 to 22.5]
Statistical Analysis 2: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Mixed Models Analysis; Geometric Mean Ratio (APL-130277/APOKYN) = 16.7, 90% CI 2-sided [13.0 to 21.3]
Statistical Analysis 3: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; Geometric Mean Ratio (APOKYN/APO-go) = 96.9, 90% CI 2-sided [74.2 to 126.4]
Statistical Analysis 4: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Ratio = 0.32 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 20 mg and APO-Go 3 mg
Statistical Analysis 5: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; Ratio = 0.16 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 20 mg and APOKYN 3 mg
Statistical Analysis 6: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; Ratio = 1.09 — The comparative bioavailability calculated as the ratio of the Test/Reference between APO-Go 3 mg and APOKYN 3 mg
Statistical Analysis 7: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Ratio = 0.23 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 25 mg and APO-Go 4 mg
Statistical Analysis 8: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; Ratio = 0.23 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 25 mg and APOKYN 4 mg
Statistical Analysis 9: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; Ratio = 1.00 — The comparative bioavailability calculated as the ratio of the Test/Reference between APO-Go 4 mg and APOKYN 4 mg
Statistical Analysis 10: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Ratio = 0.15 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 30 mg and APO-Go 5 mg
Statistical Analysis 11: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; Ratio = 0.14 — The comparative bioavailability calculated as the ratio of the Test/Reference between APL 30 mg and APOKYN 5 mg
Statistical Analysis 12: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; Ratio = 0.96 — The comparative bioavailability calculated as the ratio of the Test/Reference between APO-Go 5 mg and APOKYN 5 mg

4. Primary Outcome: Area Under the Concentration- Time Curve (AUC Inf)
Description: area under the concentration-time curve from time zero extrapolated to infinity using the linear up log down trapezoidal rule.
Time Frame: Day 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: (hxng/mL)/(mg)
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 7 | 8
(hxng/mL)/(mg) | 0.52 [0.36 to 0.76] | 2.97 [2.01 to 4.39] | 3.04 [2.08 to 4.45]
Statistical Analysis 1: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio (APL-130277/APOKYN) = 17.6, 90% CI 2-sided [13.7 to 22.5]
Statistical Analysis 2: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; Mixed Models Analysis; Geometric Mean Ratio (APL-130277/APO-go) = 17.2, 90% CI 2-sided [13.7 to 21.6]
Statistical Analysis 3: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; Mixed Models Analysis; Geometric Mean Ratio (APOKYN/APO-go) = 97.8, 90% CI 2-sided [76.6 to 124.8]

5. Primary Outcome: Mean Residence Time (MRT)
Description: Mean residence time during one dosing interval calculated using the following equation: MRT = AUMCinf/AUC inf. AUMCinf is the area under the first moment (time.plasma concentration vs. time) curve.
Time Frame: Day 1
Population: MRT was summarized by dose level
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 6 | 7
h
  APL 20 mg, APOKYN 3 mg, and APO-go 3 mg: number analyzed (Participants) | 3 | 2 | 2
  APL 20 mg, APOKYN 3 mg, and APO-go 3 mg | 1.69 (5.2) | 1.44 (4.3) | 1.21 (19.3)
  APL 25 mg, APOKYN 4 mg, and APO-go 4 mg: number analyzed (Participants) | 2 | 2 | 2
  APL 25 mg, APOKYN 4 mg, and APO-go 4 mg | 1.83 (41.5) | 1.70 (13.8) | 1.51 (19.0)
  APL 30 mg, APOKYN 5 mg, and APO-go 5 mg: number analyzed (Participants) | 3 | 2 | 3
  APL 30 mg, APOKYN 5 mg, and APO-go 5 mg | 2.15 (15.9) | 1.23 (3.4) | 1.08 (35.4)

6. Primary Outcome: Metabolite/Parent (M/P) Drug Concentration Ratio -Cmax
Description: Metabolite (apomorphine sulfate) to Parent exposure ratio, Cmax, corrected for molecular weight differences.
Time Frame: Day 1
Population: Metabolite/Parent Cmax summarized by dose level
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: no unit
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 6 | 7
no unit
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg: number analyzed (Participants) | 3 | 2 | 2
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg | 61.6 (28.8) | 15.2 (48.9) | 11.5 (4.0)
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg: number analyzed (Participants) | 2 | 2 | 2
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg | 32.0 (157.1) | 9.0 (149.3) | 7.1 (240.3)
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg: number analyzed (Participants) | 3 | 2 | 3
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg | 61.2 (87.0) | 13.7 (8.2) | 11.3 (47.6)

7. Primary Outcome: Apparent Total Clearance of the Drug From Plasma After Oral Administration (CL/F)
Description: Apparent total clearance of the drug from plasma extravascular administration, calculated as Dose/AUCinf.
Time Frame: Day 1
Population: CL/F summarized by dose level
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 6 | 7
L/h
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg: number analyzed (Participants) | 3 | 2 | 2
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg | 2766.9 (52.4) | 407.9 (33.3) | 375.6 (32.2)
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg: number analyzed (Participants) | 2 | 2 | 2
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg | 1097.8 (99.5) | 250.2 (140.6) | 253.7 (169.6)
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg: number analyzed (Participants) | 3 | 2 | 3
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg | 1952.1 (44.3) | 350.6 (4.0) | 299.2 (41.0)

8. Primary Outcome: Apparent Volume of Distribution After Non-intravenous Administration (V/F)
Description: Apparent volume of distribution after extravascular administration, calculated as Dose/(AUCinf * λz).
Time Frame: Day 1
Population: V/F summarized by dose level
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 8 | 7
L
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg: number analyzed (Participants) | 3 | 3 | 2
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg | 4440.2 (72.0) | 577.5 (44.3) | 469.3 (19.1)
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg: number analyzed (Participants) | 2 | 2 | 2
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg | 1733.4 (52.8) | 420.8 (193.7) | 372.2 (231.1)
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg: number analyzed (Participants) | 3 | 2 | 3
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg | 3419.5 (67.4) | 452.0 (14.7) | 324.2 (73.7)

9. Primary Outcome: Terminal-phase Half-life (t½)
Description: Terminal phase half-life, as calculated by the following equation: t½ = ln(2)/λz.
Time Frame: Day 1
Population: Terminal-phase half-life summarized by dose level
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 8 | 7
h
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg: number analyzed (Participants) | 3 | 2 | 2
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg | 1.11 (15.6) | 0.98 (9.9) | 0.87 (12.6)
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg: number analyzed (Participants) | 2 | 2 | 2
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg | 1.09 (34.3) | 1.17 (20.6) | 1.02 (19.7)
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg: number analyzed (Participants) | 3 | 2 | 3
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg | 1.21 (20.5) | 0.89 (18.7) | 0.75 (35.5)
Statistical Analysis 1: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APO-go; Test type: Other; p = 0.0313, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: APL-130277, Sublingual Thin Film vs Subcutaneous APOKYN; Test type: Other; p = 0.0625, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Subcutaneous APOKYN vs Subcutaneous APO-go; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Terminal-phase Rate Constant ( λz)
Description: Apparent terminal elimination rate constant, determined by log linear regression of the plasma concentration versus time data that was judged to be in the log-linear elimination phase. At least 3 data points in the terminal phase will be used in the determination of the rate constant.
Time Frame: Day 1
Population: terminal-phase rate constant summarized by dose level
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /h
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 6 | 7
/h
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg: number analyzed (Participants) | 3 | 2 | 2
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg | 0.62 (15.6) | 0.71 (9.9) | 0.80 (12.6)
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg: number analyzed (Participants) | 2 | 2 | 2
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg | 0.63 (34.3) | 0.59 (20.6) | 0.68 (19.7)
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg: number analyzed (Participants) | 3 | 2 | 3
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg | 0.57 (20.5) | 0.78 (18.7) | 0.92 (35.5)

11. Primary Outcome: Metabolite/Parent (M/P) Drug Concentration Ratio -AUC Last
Description: Metabolite (apomorphine sulfate) to Parent exposure ratio, AUClast, corrected for molecular weight differences.
Time Frame: Day 1
Population: Metabolite/Parent (M/P) drug concentration Ratio -AUC last summarized by dose level
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: no unit
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
Number analyzed (Participants) | 8 | 8 | 7
no unit
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg: number analyzed (Participants) | 3 | 2 | 2
  APL 20 mg, APOKYN 3 mg and APO-go 3 mg | 98.16 (6.4) | 36.22 (3.0) | 32.19 (9.9)
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg: number analyzed (Participants) | 2 | 2 | 2
  APL 25 mg, APOKYN 4 mg and APO-go 4 mg | 45.79 (169.9) | 18.70 (162.8) | 16.27 (221.6)
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg: number analyzed (Participants) | 3 | 2 | 3
  APL 30 mg, APOKYN 5 mg and APO-go 5 mg | 98.07 (55.4) | 33.63 (6.2) | 26.22 (43.6)

ADVERSE EVENTS:
Time Frame: 16 days
Arm/Group | APL-130277, Sublingual Thin Film | Subcutaneous APOKYN | Subcutaneous APO-go
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/7 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277, Sublingual Thin Film (N=8) | Subcutaneous APOKYN (N=7) | Subcutaneous APO-go (N=8)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277, Sublingual Thin Film (N=8) | Subcutaneous APOKYN (N=7) | Subcutaneous APO-go (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT03292016/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT03292016/SAP_001.pdf